CLINICAL TRIAL: NCT00049595
Title: BEACOPP (4 Cycles Escalated + 4 Cycles Baseline) Versus ABVD (8 Cycles) In Stage III & IV Hodgkin's Lymphoma
Brief Title: Comparison of Two Combination Chemotherapy Regimens in Treating Patients With Stage III or Stage IV Hodgkin's Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Lymphoma Trials Office (Other); Lymphoma Study Association (Other); Grup per l'Estudi dels Limfomes de Catalunya i Balears (Other); NCIC Clinical Trials Group (Network); Australasian Leukaemia and Lymphoma Group (Other); Nordic Lymphoma Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-20012; EORTC-20012 (Other: EORTC); GELA-EORTC-20012 (Other: GELA); BNLI-EORTC-20012 (Other: BNLI); GELCAB-EORTC-20012 (Other: GELCAB); NORDICLG-EORTC-20012 (Other: NLG); CAN-NCIC-EORTC-20012 (Other: NCIC CTG); ALLG-HD04 (Other: ALLG); 2004-001558-10 (EudraCT Number)
Record Dates: First submitted 2002-11-12; First posted 2003-01-27 (Estimated); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Lymphoma
Keywords: adult lymphocyte depletion Hodgkin lymphoma; adult mixed cellularity Hodgkin lymphoma; adult nodular sclerosis Hodgkin lymphoma; stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease | interventions — Bleomycin; Filgrastim; pegfilgrastim; ABVD protocol; Cyclophosphamide; Dacarbazine; Doxorubicin; Etoposide; Prednisone; Procarbazine; Vinblastine; Vincristine

ARMS (2):
- ABVD (Active Comparator): 8 cycles of ABVD
  Interventions: Biological: bleomycin sulfate; Drug: ABVD regimen; Drug: dacarbazine; Drug: doxorubicin hydrochloride; Drug: vinblastine sulfate
- BEACOPP (Experimental): 4 cycles of BEACOPP Escalated + 4 cycles of BEACOPP Baseline
  Interventions: Biological: bleomycin sulfate; Biological: filgrastim; Biological: pegfilgrastim; Drug: BEACOPP regimen; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: prednisone; Drug: procarbazine hydrochloride; Drug: vincristine sulfate

INTERVENTIONS:
Biological: bleomycin sulfate
Biological: filgrastim
  Arms: BEACOPP
Biological: pegfilgrastim
  Arms: BEACOPP
Drug: ABVD regimen
  Arms: ABVD
Drug: BEACOPP regimen
  Arms: BEACOPP
Drug: cyclophosphamide
  Arms: BEACOPP
Drug: dacarbazine
  Arms: ABVD
Drug: doxorubicin hydrochloride
Drug: etoposide
  Arms: BEACOPP
Drug: prednisone
  Arms: BEACOPP
Drug: procarbazine hydrochloride
  Arms: BEACOPP
Drug: vinblastine sulfate
  Arms: ABVD
Drug: vincristine sulfate
  Arms: BEACOPP

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells. It is not yet known which combination chemotherapy regimen is more effective in treating stage III or stage IV Hodgkin's lymphoma.

PURPOSE: Randomized phase III trial to compare the effectiveness of two combination chemotherapy regimens in treating patients who have stage III or stage IV Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare event-free survival of patients with stage III or IV Hodgkin's lymphoma treated with bleomycin, etoposide, doxorubicin, cyclophosphamide, vincristine, procarbazine, and prednisone vs doxorubicin, bleomycin, vinblastine, and dacarbazine.
* Compare complete response, disease-free survival, and overall survival of patients treated with these regimens.
* Compare quality of life of patients treated with these regimens.
* Compare occurrence of second malignancies in patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to International Prognostic Score (3 vs 4 or more) and participating center. Patients are randomized to 1 of 2 treatment arms.

* Arm I (BEACOPP): Patients receive doxorubicin IV over 5 minutes and cyclophosphamide IV on day 1; etoposide IV over 30 minutes on days 1-3; oral procarbazine on days 1-7; oral prednisone on days 1-14; and vincristine IV and bleomycin IV or intramuscularly (IM) on day 8. Patients may receive dexamethasone in place of prednisone. Patients also receive filgrastim (G-CSF) subcutaneously (SC) beginning on day 9 and continuing until blood counts recover or pegfilgrastim SC on day 9 only. Treatment repeats every 22 days for 8 courses (4 courses escalated dose followed by 4 courses baseline dose) in the absence of disease progression or unacceptable toxicity.
* Arm II (ABVD): Patients receive doxorubicin IV over 5 minutes, bleomycin IV or IM, vinblastine IV, and dacarbazine IV over 5-10 minutes on days 1 and 15. Treatment repeats every 28 days for 8 courses in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, at the end of therapy, and then annually for 10 years.

Patients are followed every 3 months for 3 years, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 550 patients (225 per treatment arm) will be accrued for this study within 5.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed Hodgkin's lymphoma

  * No lymphocyte predominant, nodular type (nodular paragranuloma)
  * Clinical stage III or IV disease
* At least 1 bidimensionally measurable target lesion or extranodal lesion
* International Prognostic Score of at least 3

PATIENT CHARACTERISTICS:

Age

* 16 to 60

Performance status

* WHO 0-2

Life expectancy

* Not specified

Hematopoietic

* WBC greater than 2,000/mm^3
* Platelet count greater than 100,000/mm^3

Hepatic

* No prior uncontrolled hepatitis B viral infection
* Bilirubin no greater than 2.5 times normal (unless due to Hodgkin's lymphoma)

Renal

* Creatinine no greater than 2.0 mg/dL (unless due to Hodgkin's lymphoma)

Cardiovascular

* No severe cardiac disease that would limit normal life expectancy or preclude study
* LVEF at least 50%

Pulmonary

* No severe pulmonary disease that would limit normal life expectancy or preclude study
* Respiratory function at least 30%

Other

* HIV negative
* HTLV1 negative
* No severe active infection
* No severe neurological or metabolic disease that would limit normal life expectancy or preclude study
* No other prior or concurrent malignancy except basal cell skin cancer or carcinoma in situ of the cervix
* No psychological, familial, sociological, or geographical condition that would preclude study
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* No concurrent radiotherapy

Surgery

* Not specified

Other

* No prior therapy for Hodgkin's lymphoma

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 552 (Actual)
Dates: Start 2002-08 (Actual); Primary Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Event-free survival | from randomization to early discontinuation of protocol treatment, no CR/CRu after 8 cycles, relapse, progression or death

SECONDARY OUTCOMES:
Complete response as assessed by Cheson criteria adapted to Hodgkin's lymphoma | from randomization till end of treatment
Disease-free survival in patients with complete response | from the day of first documentation of CR to the day of relapse
Overall survival | from the date of randomization to the date of death
Quality of life as assessed by European Organization for Research of the Treatment of Cancer (EORTC) Quality of Life Questionnaire (QoLQ) C30 version 3.0 | from one week prior to randomization till 10 years after end of treatment or death

CONTACTS AND LOCATIONS:
Overall Officials: Patrice P. Carde, MD, Study Chair — Gustave Roussy, Cancer Campus, Grand Paris; David C. Linch, Study Chair — Middlesex Hospital; Marine Divine, MD, Study Chair — Centre Hospitalier Universitaire Henri Mondor; Anna Sureda, Study Chair — Hospital de la Santa Cruz i Sant Pau; Ralph M. Meyer, MD, FRCPC, Study Chair — Margaret and Charles Juravinski Cancer Centre; David Ma, MD, Study Chair — St Vincent's Hospital; Devinder Gill, MD, Study Chair — Princess Alexandra Hospital; Bengt Glimelius, MD, Study Chair — Uppsala University Hospital
Locations (140):
- Australia (7):
  - Canberra Hospital, Garran, Australian Capital Territory
  - Nepean Cancer Care Centre at Nepean Hospital, Kingswood, New South Wales
  - Westmead Institute for Cancer Research at Westmead Hospital, Westmead, New South Wales
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Peter MacCallum Cancer Centre, East Melbourne, Victoria
  - St. Vincent's Hospital - Melbourne, Fitzroy, Victoria
  - Royal Perth Hospital, Perth, Western Australia
- Belgium (14):
  - Ziekenhuis Netwerk Antwerpen Middelheim, Antwerp
  - AZ Sint-Jan, Bruges
  - Institut Jules Bordet, Brussels
  - Hopital Universitaire Erasme, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - Centre Hospitalier Universitaire Brugmann, Brussels
  - Centre Hospitalier Notre Dame - Reine Fabiola, Charleroi
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Algemeen Ziekenhuis Sint Lucas, Ghent
  - Hopital de Jolimont, Haine-Saint-Paul
  - U.Z. Gasthuisberg, Leuven
  - Centre Hospitalier Regional de la Citadelle, Liège
  - H. Hartziekenhuis - Roeselaere, Roeselare
  - Clinique Universitaire De Mont-Godinne, Yvoir
- Canada (22):
  - Tom Baker Cancer Centre - Calgary, Calgary, Alberta
  - Cross Cancer Institute at University of Alberta, Edmonton, Alberta
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Centre Hospitalier De Dunkerque - CHD, Winnipeg, Manitoba
  - Moncton Hospital, Moncton, New Brunswick
  - Doctor H. Bliss Murphy Cancer Centre, St. John's, Newfoundland and Labrador
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - Northeastern Ontario Regional Cancer Centre, Greater Sudbury, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston General Hospital, Kingston, Ontario
  - London Regional Cancer Program at London Health Sciences Centre, London, Ontario
  - Ottawa Hospital Regional Cancer Centre - General Campus, Ottawa, Ontario
  - Edmond Odette Cancer Centre at Sunnybrook, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Windsor Regional Cancer Centre at Windsor Regional Hospital, Windsor, Ontario
  - Hopital Charles Lemoyne, Greenfield Park, Quebec
  - Maisonneuve-Rosemont Hospital, Montreal, Quebec
  - Hopital Notre-Dame du CHUM, Montreal, Quebec
  - CHUM - Hotel Dieu Hospital, Montreal, Quebec
  - McGill Cancer Centre at McGill University, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Québec, Quebec
  - Hopital du Saint-Sacrement - Quebec, Québec, Quebec
  - Saskatoon Cancer Centre at the University of Saskatchewan, Saskatoon, Saskatchewan
- University Hospital Rebro, Zagreb, Croatia
- Thomayer's University Hospital, Prague, Czechia
- France (55):
  - Centre Hospitalier d'Annecy, Annecy
  - Centre Hospitalier de la Cote Basque, Bayonne
  - Centre Hospitalier Regional de Besancon - Hopital Jean Minjoz, Besançon
  - Institut Bergonie, Bordeaux
  - Polyclinique Bordeaux Nord Aquitaine, Boucher
  - C.H. Bourg En Bresse, Bourg-en-Bresse
  - CHU de Caen, Caen
  - Polyclinique Du Parc, Caen
  - Centre Regional Francois Baclesse, Caen
  - Centre Hospitalier Regional de Chambery, Chambéry
  - Hopital d'Instruction des Armees Percy, Clamart
  - Hopital Antoine Beclere, Clamart
  - CHR Clermont Ferrand, Hotel Dieu, Clermont-Ferrand
  - Hopital Louis Pasteur, Colmar
  - Centre Hospitalier Sud Francilien - Site Corbeil, Corbeil
  - Centre Hospitalier Universitaire Henri Mondor, Créteil
  - Hopital Du Bocage, Dijon
  - Institut Prive de Cancerologie, Grenoble
  - Hopital Andre Mignot, Le Chesnay
  - Hopital Saint Antoine Lille, Lille
  - Centre Hospitalier Regional et Universitaire de Lille, Lille
  - Centre Hospital Regional Universitaire de Limoges, Limoges
  - Centre Leon Berard, Lyon
  - Hopital Edouard Herriot - Lyon, Lyon
  - Marseille Institute of Cancer - Institut J. Paoli and I. Calmettes, Marseille
  - Centre Hospitalier de Meaux, Meaux
  - Centre Hospitalier Marc Jacquet, Melun
  - Hopital Notre-Dame de Bon Secours, Metz
  - Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier
  - Centre Hospitalier de Mulhouse, Mulhouse
  - Centre Antoine Lacassagne, Nice
  - Hopital de l'Archet CHU de Nice, Nice
  - Hotel Dieu de Paris, Paris
  - Institut Curie Hopital, Paris
  - Hopital Saint-Louis, Paris
  - Hopital Saint Antoine, Paris
  - CHU Pitie-Salpetriere, Paris
  - Hopital Cochin, Paris
  - Hopital Necker, Paris
  - Hopital Haut Leveque, Pessac
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Hopital Rene Dubos, Pontoise
  - Institut Jean Godinot, Reims
  - Hopital Sud, Rennes
  - Centre Henri Becquerel, Rouen
  - Centre Rene Huguenin, Saint-Cloud
  - CHU Sainte-Etienne - Hopital Bellevue, Saint-Etienne
  - Hopital de Saint Germain-en-Laye, Saint-Germain-en-Laye
  - Hopital Universitaire Hautepierre, Strasbourg
  - Hopital Foch, Suresnes
  - Centre Hospitalier Valence, Valence
  - Centre Hospitalier de Valenciennes, Valenciennes
  - CHU de Nancy - Hopitaux de Brabois, Vandœuvre-lès-Nancy
  - Hopital Paul Brousse, Villejuif
  - Institut Gustave Roussy, Villejuif
- National Institute of Oncology, Budapest, Hungary
- Netherlands (16):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Meander Medisch Centrum, Amersfoort
  - Netherlands Cancer Institute - Antoni van Leeuwenhoek Hospital, Amsterdam
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Academisch Medisch Centrum at University of Amsterdam, Amsterdam
  - Reinier de Graaf Group - Delft, Delft
  - Medisch Spectrum Twente, Enschede
  - University Medical Center Groningen, Groningen
  - Atrium Medical Centre - Heerlen, Heerlen
  - Leiden University Medical Center, Leiden
  - Academisch Ziekenhuis Maastricht, Maastricht
  - Universitair Medisch Centrum St. Radboud - Nijmegen, Nijmegen
  - Saint Laurentius Ziekenhuis, Roermond
  - Daniel Den Hoed Cancer Center at Erasmus Medical Center, Rotterdam
  - HagaZiekenhuis - Locatie Leyenburg, The Hague
  - University Medical Center Utrecht, Utrecht
- New Zealand (2):
  - Auckland City Hospital, Auckland
  - Waikato Hospital, Hamilton
- Maria Sklodowska-Curie Memorial Cancer Center and Institute of Oncology - Warsaw, Warsaw, Poland
- Spain (3):
  - Hospital de la Santa Cruz i Sant Pau, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitari Germans Trias i Pujol, Barcelona
- Sweden (6):
  - Sahlgrenska University Hospital, Gothenburg (Goteborg)
  - University Hospital of Linkoping, Linköping
  - Lund University Hospital, Lund
  - Karolinska University Hospital - Huddinge, Stockholm
  - Umea Universitet, Umeå
  - Uppsala University Hospital, Uppsala
- United Kingdom (11):
  - Queen Elizabeth Hospital at University Hospital of Birmingham NHS Trust, Birmingham, England
  - Raigmore Hospital, Birmingham, England
  - Kent and Canterbury Hospital, Canterbury, England
  - Hull Royal Infirmary, Hull, England
  - Kettering General Hosptial, Kettering, England
  - Leicester Royal Infirmary, Leicester, England
  - Middlesex Hospital, London, England
  - Mount Vernon Cancer Centre at Mount Vernon Hospital, Northwood, England
  - Nottingham City Hospital NHS Trust, Nottingham, England
  - Cancer Research Centre at Weston Park Hospital, Sheffield, England
  - Staffordshire General Hospital, Stafford, England

REFERENCES:
- [Derived] Carde P, Karrasch M, Fortpied C, Brice P, Khaled H, Casasnovas O, Caillot D, Gaillard I, Bologna S, Ferme C, Lugtenburg PJ, Morschhauser F, Aurer I, Coiffier B, Meyer R, Seftel M, Wolf M, Glimelius B, Sureda A, Mounier N. Eight Cycles of ABVD Versus Four Cycles of BEACOPPescalated Plus Four Cycles of BEACOPPbaseline in Stage III to IV, International Prognostic Score >/= 3, High-Risk Hodgkin Lymphoma: First Results of the Phase III EORTC 20012 Intergroup Trial. J Clin Oncol. 2016 Jun 10;34(17):2028-36. doi: 10.1200/JCO.2015.64.5648. Epub 2016 Apr 25. PMID 27114593